CLINICAL TRIAL: NCT01220414
Title: Attenuation of Pain in Men and Women: Mechanisms of Exercise-Induced Analgesia
Brief Title: Attenuation of Pain in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-2010-0087
Record Dates: First submitted 2010-09-28; First posted 2010-10-13 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Men (Active Comparator)
  Interventions: Drug: Naltrexone, then placebo; Drug: Placebo, then Naltrexone
- Women (Active Comparator)
  Interventions: Drug: Naltrexone, then placebo; Drug: Placebo, then Naltrexone

INTERVENTIONS:
Drug: Naltrexone, then placebo — 50 mg of naltrexone
Drug: Placebo, then Naltrexone — sugar pill

SUMMARY:
The purpose of this study is to examine opioid and endocannabinoid mechanisms of exercise-induced analgesia in men and women.

ELIGIBILITY:
Inclusion Criteria: Healthy men and women

-

Exclusion Criteria:

* current cardiac or other chronic diseases (e.g., cancer, diabetes, hypertension, kidney disease); routine use of prescriptive medications; history of vasovagal response to phlebotomy; an allergy to naltrexone; pregnancy; current smokers; current use of recreational drugs; history of substance abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Males, Naltrexone Then Placebo | Males, Placebo Then Naltrexone | Females, Naltrexone Then Placebo | Females, Placebo Then Naltrexone
Started | 15 | 14 | 14 | 15
Completed | 14 | 14 | 14 | 14
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Naltrexone Then Placebo: All participants completed both naltrexone and placebo conditions
- Total: Total of all reporting groups
Arm/Group | Naltrexone Then Placebo | Placebo Then Naltrxone | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (3) | 21 (3) | 21 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Time for Subject to Reach Pain Threshold
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Men, Placebo | Women, Placebo | Men, Naltrexone | Females, Naltrexone
Number analyzed (Participants) | 14 | 15 | 15 | 14
seconds
  Pain threshold at baseline | 16.1 (12.1) | 16.0 (24.0) | 15.0 (10.0) | 14.8 (24.0)
  Pain threshold post exercise | 28.8 (27.6) | 24.1 (35.3) | 28.4 (26.6) | 22.5 (30.1)

ADVERSE EVENTS:
Groups:
- Naltrexone and Placebo: Participants completed both naltrexone and placebo conditions
Arm/Group | Naltrexone and Placebo
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No